CLINICAL TRIAL: NCT00923793
Title: Comparison of Individual CAD/CAM-based Implants Consisting on Hydroxylapatite and Titanium to be Used in Cranioplasty - a Randomized Multicenter Clinical Trial
Brief Title: Comparison of Individual Computer Aided Design/Manufactured (CAD/CAM) - Based Implants Consisting on Hydroxylapatite and Titanium to be Used in Cranioplasty
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was stopped, due to slow recruitment rate
Sponsor: University of Leipzig (Other)
Collaborators: Universitätsklinikum Leipzig (Other)
Responsible Party: Principal Investigator, Dirk Lindner, Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CustomBone vs. Titanium
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Skull Defects; Cranioplasty
Keywords: skull defects; Hydroxylapatite implant; Titanium implant; calotte defects without the possibility to be covered with the missing own bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titanium (Active Comparator): Titanium implant for cranioplasty. Titanium implants are used since 10 years in Germany because of their high biocompatibility and accuracy of fit.
  Interventions: Device: Titanium implant (CranioConstruct™)
- Hydroxylapatite (Experimental): Hydroxylapatite (CustomBone) implant Hydroxylapatite implants are used since about 3 years in Germany. As this material is very similar to human bone structure an improved osteointegration has been observed.
  Interventions: Device: Hydroxylapatite (CustomBone)

INTERVENTIONS:
Device: Titanium implant (CranioConstruct™) — One to three weeks before operation the skull defect is well defined using Computer tomography. Based on these results the Titanium implant is ordered.
  Other Names: CranioConstruct™
  Arms: Titanium
Device: Hydroxylapatite (CustomBone) — Six to eight weeks before operation the skull defect is well defined using Computer tomography. Based on these results the Hydroxylapatite implant is ordered.
  Other Names: CustomBone
  Arms: Hydroxylapatite

SUMMARY:
The purpose of this study is to compare the results of cranioplasty with CAD/CAM (computer aided design/manufactured) based Hydroxylapatite and Titanium implants in respect to infections, re-operations, antibiotic treatment or removal of the implant.

DETAILED DESCRIPTION:
Both implant materials for cranioplasty, Hydroxylapatite and Titanium, are CE certified medical devices used in common practices. This study is intended to get prospective data in addition to the empirical and retrospective existing ones to enable the decision on which implant material should be preferably employed in future.

ELIGIBILITY:
Inclusion Criteria:

1. Skull defects without the possibility to be covered with the missing own bone
2. Size of the defect ≥ 16 cm2
3. Age ≥ 18
4. Written informed consent of the patient

Exclusion Criteria:

1. Active tumor
2. ASA 4 classification
3. Allergic disposition to ceramic or titanium
4. Concomitant participation in other clinical trials
5. Pregnant or nursing women
6. Expected low compliance
7. HIV positive
8. Active drug abuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of local and/or systemic infections (acute/chronic) in both study arms within the first 6 months after operation. | 6 months

SECONDARY OUTCOMES:
Comparison of the rate of re-operations with and without ex-plantation of the implant in both arms. | 6 months
Comparison of post-operative computer tomography (CT) (native and bone 5 mm) within 48 h in respect to bleeding, dislocation and further complications after cranioplasty in both arms. | 48 hours post-operative
Comparison of health-related quality of life after cranioplasty in both arms using the SF36-questionnaire. | 6 months
Comparison between both groups referring to cosmetic result, period of hospitalization, costs, intra-operative features. | 6 months
Comparison of temperature sensitivity (cold/heat) six months after implantation in both groups. | 6 months
Description of osteointegration with CT and bone scan six months post-operative in both groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Lindner, Dr. med., Study Director — Universität Leipzig KöR Medizinische Falkutät Klinif für Neurochirurgie
Locations (1):
- Universität Leipzig KöR Medizinische Fakultät Klinik für Neurochirurgie, Leipzig, Saxony, Germany

REFERENCES:
- [Background] Eufinger H, Weihe S, Scherer P, Rasche C, Wehmöller M. Management of cranial and craniofacial bone defects with prefabricated individual titanium implants: follow-up and evaluation of 166 patients with 169 titanium implants from 1994 to 2000. Int. J. CARS 2006; 1: 197-203
- [Derived] Lindner D, Schlothofer-Schumann K, Kern BC, Marx O, Muns A, Meixensberger J. Cranioplasty using custom-made hydroxyapatite versus titanium: a randomized clinical trial. J Neurosurg. 2017 Jan;126(1):175-183. doi: 10.3171/2015.10.JNS151245. Epub 2016 Feb 26. PMID 26918471